CLINICAL TRIAL: NCT01072994
Title: Fish Oil Effect on Heart Muscle Cells in Heart Transplant Patients (FOHMC)
Brief Title: Fish Oil In Heart Transplantation
Acronym: FOHMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Mandeep R. Mehra, Professor and Head of Cardiology, University of Maryland School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 691; P20HL101434 (NIH)
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2010-02

CONDITIONS: Myocardial Tissue in Heart Transplantation
Keywords: Myocardium; Phospholipid; Fish oil; Cardiolipin; Transplantation
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Fish Oil — Differential proportional doses of DHA versus DHA and EPA

SUMMARY:
Despite aggressive treatment, patients with heart failure have a poor prognosis. Docosahexaenoic acid (DHA), an omega-3 polyunsaturated fatty acids found in fish oils, may prevent the progressions of heart failure through mechanisms that are not addressed with current drugs.

The omega-3 polyunsaturated fatty acids Docosahexaenoic Acid (DHA) and Eicosapentaenoic acid (EPA) favorably impact mitochondrial dysfunction and chronic inflammation in heart failure (HF). Treatment with DHA-t-EPA alters cardiac phospholipid composition by decreasing arachidonic acid (a pro-inflammatory fatty acid) and increasing DHA and the mitochondrial phospholipid cardiolipin, with is associated with improved Left Ventricular (LV) function.

Fish oil supplements contain a mix of DHA and EPA, however we postulate that DHA is superior to EPA in improving mitochondrial function and suppressing inflammation, and thus DHA should be used to treat HF.

Cardiac phospholipid fatty acid composition (i.e. DHA, EPA, and arachidonic acid) and cardiolipin (CL) content will be measured in biopsies from stable heart transplantation patients that are obtained as part of standard clinical care in heart transplant patients before and after treatment with DHA alone or DHA+EPA. We will compare cardiac phospholipid composition from biopsies obtained at study entry and at 6 months follow-up (allowable range +/- two months, depending on patients' clinical conditions).

DETAILED DESCRIPTION:
50 adult heart transplant recipients (18-75 years of age) entered the maintenance phase (>6 months after heart transplantation), remaining clinically quiescent (See Inclusion criteria) and undergoing regularly scheduled myocardial biopsies (as part of standard clinical care) for allograft rejection will be recruited.

Half of the subject will be receive DHA and half DHA+EPA administered orally which will be administered in two capsules in the morning and two in the evening. Each patient will serve as their own control, and comparisons will be made between pre and post treatments within each patient.

Prior to assignment to treatment, a septal biopsy (10 to 20 mg) will be obtained during a routine biopsy procedure and immediately frozen in liquid nitrogen and stored at -80 until analysis. Therapy will continue for at least 6 months and until completion of the primary end point of paired cardiac biopsy acquisition. Cardiac biopsies obtained during regularly scheduled myocardial biopsies for clinical evaluation for allograft rejection will also be analyzed for phospholipid fatty acid composition.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years of age at time of cardiac transplantation;
2. Absence of cardiac allograft rejection on the index cardiac biopsy
3. No treatment for cardiac allograft rejection within 30 days of enrollment
4. Absence of restrictive physiology or cardiac allograft dysfunction on hemodynamic assessment
5. Stable immunosuppression and other background medications for past 30 days with no planned modulation in therapy for 6 months
6. All women of childbearing potential must have a negative urine pregnancy test prior to treatment and agree to use adequate contraception (defined as oral or injectable contraceptives, intrauterine devices, surgical sterilization or a combination of a condom and spermicide) or limit sexual activity to vasectomized partner for 3 months after administration of therapy;
7. Ability to sign Informed Consent Form and Release of Medical Information Form

Exclusion Criteria:

1. Regular use of u)-3 PUFA supplements (fish oil or flax seed oil).
2. Alcoholism or drug abuse;
3. Poorly controlled diabetes (defined as a Hb A1C >8);
4. Fasting triglycerides >250 mg/dl.
5. Pregnancy and Lactation
6. Persons with known sensitivity or allergy to fish;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Cardiac phospholipid fatty acid composition and cardiolipin (CL) content in myocardium | 6 months
  Cardiac phospholipid fatty acid composition (i.e. DHA, EPA, and arachidonic acid) and cardiolipin (CL) content will be measured in biopsies from stable heart transplantation patients that are obtained as part of standard clinical care before and after treatment with DHA alone or DHA+EPA. We will compare cardiac phospholipid composition from biopsies obtained at study entry and at 6 months follow-up (allowable range +/- two months, depending on patients' clinical schedule).